CLINICAL TRIAL: NCT05131230
Title: A Prospective, Multi-Centre, Propensity Score Based Matched Pair Controlled, Study of Standard Medical Care Plus CytoSorb® 300 mL Device Compared to Standard Medical Care Alone in Patients With Acute on Chronic Liver Failure Due to Severe Alcoholic Hepatitis in Combination With Systemic Hyperinflammation and Acute on Chronic Liver Failure Score ≥2
Brief Title: CytoSorb® in Patients With Acute on Chronic Liver Failure
Acronym: HepOnFire
Status: Withdrawn | Type: Observational
Why Stopped: No patients enrolled
Sponsor: CytoSorbents Europe GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: L02HOF
Record Dates: First submitted 2021-11-12; First posted 2021-11-23 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Acute on Chronic Liver Failure; Alcoholic Hepatitis
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; Hepatitis, Alcoholic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CytoSorb group
  Interventions: Device: CytoSorb® treatment

INTERVENTIONS:
Device: CytoSorb® treatment — Patients with Acute on Chronic Liver Failure (ACLF) due to Severe Alcoholic Hepatitis in combination with systemic inflammation and ACLF grade ≥2 will be enrolled in this study. Every patient that is screened, fulfills the inclusion/exclusion criteria, and consents to the study, will be allowed to enter the study. Patients will receive Standard of Care treatment for alcoholic hepatitis plus treatment with the CytoSorb® 300 mL device.

SUMMARY:
The objective of this study is to assess the safety and performance of the CytoSorb® therapy in patients with Acute on Chronic Liver Failure (ACLF) grade ≥ 2 due to a severe alcohol induced hepatitis (Maddrey DF > 32) and a severe inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18
2. Signed Informed Consent Form (ICF)
3. Total bilirubin ≥ 8 mg/dL
4. Acute Alcoholic Hepatitis diagnosed by EtOH consumption within 6 weeks of onset of symptoms, exclusion of other causes for jaundice and liver biopsy or at least 2 out of the following symptoms:

   * Hepatomegaly
   * AST > ALT
   * Elevated WBC
   * Ascites
5. Maddrey DF > 32
6. Systemic inflammation as defined by 2 fulfilled criteria out of:

   * leucocytosis
   * body temperature > 38°C
   * tachycardia > 90 bpm
   * tachypnoeia > 20 breaths/min
7. ACLF grade ≥2
8. Creatinine >2 mg/dl and increase >1.5 mg/dl despite standard of care

Exclusion Criteria:

1. Platelets < 40,000/mm3
2. INR > 3.5
3. MELD Score > 35
4. AST > 500 IU/l
5. Bilirubin reduction > 20% in prior 72 hours (early responders to conventional Standard of Care (SOC))
6. Uncontrolled infection, bleeding or hemodynamic instability
7. Small liver size (diagnosed by imaging, ultrasound/CT)
8. Chronic dialysis
9. Contraindications for CytoSorb® according to Instructions for Use
10. ACLF grade <2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 patients meeting the eligibility requirements of the study will receive Standard of Care treatment for alcoholic hepatitis (including steroid therapy according to AASLD/EASL guidelines and extracorporeal treatments when indicated) plus treatment with the CytoSorb® 300 mL device, a hemoperfusion adsorbent CE-certified therapy for the removal of bilirubin and pro-inflammatory cytokines (CytoSorb group).
  30 propensity score matched controls from a patient database will be drawn from existing US and European sources (prospectively collected databases from geographies with comparable Standard of Care). The 30 CytoSorb group patients will be compared with these database patients.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients in each group with Acute on Chronic Liver Failure (ACLF) grade <2 | 7 Days
  To evaluate effectiveness of the CytoSorb® treatment compared to control group by comparing the proportion of patients in each group with ACLF grade <2 at the end of Day 7 after CytoSorb® therapy start (assessed by https://www.efclif.com/scientific-activity/score-calculators/clif-c-aclf).
Safety of CytoSorb treatment | 30 Days
  To evaluate if CytoSorb® treatment plus Standard Medical Care (SMC) compared to SMC alone is safe and tolerable as assessed by the incidence of SA(D)Es, ADEs, DDs, SADEs, and USADEs.
  SAE - Severe Adverse Effect; ADE - Adverse Device Effect; SADE - Severe Adverse Device Effect; DD - Device Deficiencies; USADE - Unexpected Serious Adverse Device Effect

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Universitätsklinikum Knappschaftskrankenhaus Bochum GmbH, Bochum
  - University of Rostock, Rostock